CLINICAL TRIAL: NCT02279641
Title: A Phase 1b, Randomized, Open-label Study to Evaluate the Potential Pharmacokinetic and Pharmacodynamic Interactions Between RDEA3170 and Allopurinol in Adult Male Subjects With Gout
Brief Title: RDEA3170 and Allopurinol Combination Study in Gout Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ardea Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RDEA3170-107
Record Dates: First submitted 2014-10-28; First posted 2014-10-31 (Estimated); Results first posted 2017-12-20 (Actual); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Gout
MeSH Terms: conditions — Gout | interventions — verinurad; Allopurinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence A (Experimental): RDEA3170 qd (once daily), RDEA3170 + allopurinol qd, allopurinol qd
  Interventions: Drug: RDEA3170 10 mg; Drug: allopurinol 300 mg
- Sequence B (Experimental): allopurinol qd, RDEA3170 + allopurinol qd, RDEA3170 qd
  Interventions: Drug: RDEA3170 10 mg; Drug: allopurinol 300 mg

INTERVENTIONS:
Drug: RDEA3170 10 mg
Drug: allopurinol 300 mg

SUMMARY:
This is a Phase 1b, randomized, open-label, drug-drug interaction study in adult male subjects with gout. It is designed to assess the pharmacokinetics (PK) and pharmacodynamics (PD) of RDEA3170 or allopurinol alone and in combination in the fed state.

ELIGIBILITY:
Inclusion Criteria:

* Subject meets one or more criteria for the diagnosis of gout as per the American Rheumatism Association Criteria for the Classification of Acute Arthritis of Primary Gout.
* Subject has a body weight ≥ 50 kg (110 lbs.) and a body mass index ≥ 18 and ≤ 45 kg/m2.
* Subject has a Screening serum urate level ≥ 8 mg/dL and ≤ 10 mg/dL
* Subject is free of any clinically significant disease or medical condition, per the Investigator's judgment.

Exclusion Criteria:

* Subject is unable to take colchicine for gout flare prophylaxis.
* Subject has a history or suspicion of kidney stones.
* Subject has an estimated creatinine clearance < 60 mL/min calculated by the Cockcroft-Gault formula using ideal body weight at Screening prior to Day -2.
* Subject is on unstable doses of chronic medications. Subjects taking medications for chronic medical conditions must be on stable doses during the course of the study, including the Screening period. Dose adjustments are allowed if deemed medically necessary by the investigator and following discussion with the medical monitor
* Chronic and stable doses of losartan, fenofibrate, guaifenesin, and sodium-glucose linked transporter-2 inhibitors are permitted if the dose is stable for at least 14 days prior to study medication dosing.
* Subject is unable or unwilling to comply with the study requirements or has a situation or condition that, in the opinion of the Investigator, may interfere with participation in the study.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2015-04-06 (Actual); Study Completion 2015-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Hall, MD, Study Director — Ardea Biosciences, Inc.
Locations (1):
- Overland Park, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 12 subjects were randomized
Pre-assignment Details: Twelve subjects were randomized to 1 of 2 treatment sequences (Sequence A or B) in a 1:1 ratio.
Groups:
- RDEA3170 or Allopurinol Alone and in Combination (Sequence A): Days 1 to 7: 10 mg once daily (qd) RDEA3170; Days 8 to 14: 10 mg qd RDEA3170 + 300 mg qd allopurinol; Days 15 to 21: 300 mg qd allopurinol
- RDEA3170 or Allopurinol Alone and in Combination (Sequence B): Days 1 to 7: 300 mg qd allopurinol; Days 8 to 14: 10 mg qd RDEA3170 + 300 mg qd allopurinol; Days 15 to 21: 10 mg qd RDEA3170
Period: Overall Study
Arm/Group | RDEA3170 or Allopurinol Alone and in Combination (Sequence A) | RDEA3170 or Allopurinol Alone and in Combination (Sequence B)
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sequence A: Days 1 to 7: 10 mg once daily (qd) RDEA3170; Days 8 to 14: 10 mg qd RDEA3170 + 300 mg qd allopurinol; Days 15 to 21: 300 mg qd allopurinol
- Sequence B: Days 1 to 7: 300 mg qd allopurinol; Days 8 to 14: 10 mg qd RDEA3170 + 300 mg qd allopurinol; Days 15 to 21: 10 mg qd RDEA3170
- Total: Total of all reporting groups
Arm/Group | Sequence A | Sequence B | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53 (10.1) | 49 (10.4) | 51 (10.0)
Age, Customized [Number; unit: Participants]
  <65 | 6 | 6 | 12
  >=65 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 6 | 12
Region of Enrollment [Number; unit: Participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: Cmax of Allopurinol/Oxypurinol Alone and In Combination with RDEA3170
Time Frame: 22 days
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Groups:
- Allopurinol: Allopurinol Alone; Oxypurinol: Allopurinol Alone: Allopurinol 300 mg qd
- Allopurinol: RDEA3170 + Allopurinol; Oxypurinol: RDEA3170 + Allopurinol: RDEA3170 10 mg qd + Allopurinol 300 mg qd
Arm/Group | Allopurinol: Allopurinol Alone | Allopurinol: RDEA3170 + Allopurinol | Oxypurinol: Allopurinol Alone | Oxypurinol: RDEA3170 + Allopurinol
Number analyzed (Participants) | 12 | 12 | 12 | 12
μg/mL | 1.13 [0.894 to 1.43] | 1.51 [1.24 to 1.82] | 12.8 [11.7 to 14.0] | 8.68 [7.99 to 9.43]
Statistical Analysis 1: Comparison: Allopurinol: Allopurinol Alone vs Allopurinol: RDEA3170 + Allopurinol; Test type: Non-Inferiority or Equivalence — Informal BE assessment using the conventional BE limits of 80% to 125%; Mixed Models Analysis; Fixed effect for treatment and random effects for subjects. GLMSRs are back-transformed to the original scale; Geometric Least Squares Mean Ratio (%) = 133, 90% CI 2-sided [111 to 159]
Statistical Analysis 2: Comparison: Oxypurinol: Allopurinol Alone vs Oxypurinol: RDEA3170 + Allopurinol; Test type: Non-Inferiority or Equivalence — Informal BE assessment using the conventional BE limits of 80% to 125%; Mixed Models Analysis; Fixed effect for treatment and random effects for subjects. GLMSRs are back-transformed to the original scale; Geometric Least Squares Mean Ratio (%) = 67.9, 90% CI 2-sided [65.2 to 70.7]

2. Primary Outcome: Time of Occurrence of Maximum Observed Concentration (Tmax)
Description: Tmax of Allopurinol/Oxypurinol and RDEA3170 Alone and In Combination
Time Frame: 22 days
Measure: Median (Full Range); unit: hr
Groups:
- RDEA3170: RDEA3170 Alone: RDEA3170 10 mg qd
- RDEA3170: RDEA3170 + Allopurinol: RDEA3170 10 mg qd + Allopurinol 300 mg qd
Arm/Group | Allopurinol: Allopurinol Alone | Allopurinol: RDEA3170 + Allopurinol | Oxypurinol: Allopurinol Alone | Oxypurinol: RDEA3170 + Allopurinol | RDEA3170: RDEA3170 Alone | RDEA3170: RDEA3170 + Allopurinol
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12
hr | 1.50 [1.00 to 4.00] | 1.25 [0.500 to 4.00] | 4.00 [1.50 to 6.00] | 3.50 [1.50 to 8.00] | 3.00 [1.50 to 4.00] | 3.00 [2.00 to 10.0]

3. Primary Outcome: Area Under the Concentration-time Curve From Time Zero up to 24 Hours Postdose (AUC 0-24)
Description: AUC 0-24 of Allopurinol/Oxypurinol Alone and In Combination with RDEA3170
Time Frame: 22 days
Measure: Geometric Mean (95% Confidence Interval); unit: μg·hr/mL
Arm/Group | Allopurinol: Allopurinol Alone | Allopurinol: RDEA3170 + Allopurinol | Oxypurinol: Allopurinol Alone | Oxypurinol: RDEA3170 + Allopurinol | RDEA3170: RDEA3170 + Allopurinol
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
μg·hr/mL | 3.69 [3.24 to 4.21] | 3.68 [3.28 to 4.13] | 255 [229 to 284] | 157 [140 to 177] | 115 [96.5 to 137]
Statistical Analysis 1: Comparison: Allopurinol: Allopurinol Alone vs Allopurinol: RDEA3170 + Allopurinol; Test type: Non-Inferiority or Equivalence — Informal BE assessment using the conventional BE limits of 80% to 125%; Mixed Models Analysis; Fixed effect for treatment and random effects for subjects. GLMSRs are back-transformed to the original scale; Geometric Least Squares Mean Ratio (%) = 102, 90% CI 2-sided [93.3 to 111]
Statistical Analysis 2: Comparison: Oxypurinol: Allopurinol Alone vs Oxypurinol: RDEA3170 + Allopurinol; Test type: Non-Inferiority or Equivalence — Informal BE assessment using the conventional BE limits of 80% to 125%; Mixed Models Analysis; Fixed effect for treatment and random effects for subjects. GLMSRs are back-transformed to the original scale; Geometric Least Squares Mean Ratio (%) = 61.8, 90% CI 2-sided [58.1 to 65.7]
Statistical Analysis 3: Comparison: RDEA3170: RDEA3170 + Allopurinol; Test type: Non-Inferiority or Equivalence — Informal BE assessment using the conventional BE limits of 80% to 125%; Mixed Models Analysis; Fixed effect for treatment and random effects for subjects. GLMSRs are back-transformed to the original scale; Geometric Least Squares Mean Ratio (%) = 95.9, 90% CI 2-sided [88.4 to 104]

4. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to the Last Quantifiable Sampling Timepoint (AUC Last)
Description: AUC last of Allopurinol/Oxypurinol Alone and In Combination with RDEA3170
Time Frame: 22 days
Measure: Geometric Mean (95% Confidence Interval); unit: μg·hr/mL
Arm/Group | Allopurinol: Allopurinol Alone | Allopurinol: RDEA3170 + Allopurinol | Oxypurinol: Allopurinol Alone | Oxypurinol: RDEA3170 + Allopurinol
Number analyzed (Participants) | 12 | 12 | 12 | 12
μg·hr/mL | 3.50 [3.04 to 4.04] | 3.61 [3.22 to 4.05] | 255 [229 to 284] | 157 [140 to 177]
Statistical Analysis 1: Comparison: Allopurinol: Allopurinol Alone vs Allopurinol: RDEA3170 + Allopurinol; Test type: Non-Inferiority or Equivalence — Informal BE assessment using the conventional BE limits of 80% to 125%; Mixed Models Analysis; Fixed effect for treatment and random effects for subjects. GLMSRs are back-transformed to the original scale; Geometric Least Squares Mean Ratio (%) = 103, 90% CI 2-sided [94.9 to 112]
Statistical Analysis 2: Comparison: Oxypurinol: Allopurinol Alone vs Oxypurinol: RDEA3170 + Allopurinol; Test type: Non-Inferiority or Equivalence — Informal BE assessment using the conventional BE limits of 80% to 125%; Mixed Models Analysis; Fixed effect for treatment and random effects for subjects. GLMSRs are back-transformed to the original scale; Geometric Least Squares Mean Ratio (%) = 61.8, 90% CI 2-sided [58.1 to 65.7]

5. Primary Outcome: Apparent Terminal Half-life (t1/2)
Description: t1/2 of Allopurinol/Oxypurinol and RDEA3170 Alone and In Combination
Time Frame: 22 days
Measure: Geometric Mean (95% Confidence Interval); unit: hr
Arm/Group | Allopurinol: Allopurinol Alone | Allopurinol: RDEA3170 + Allopurinol | Oxypurinol: Allopurinol Alone | Oxypurinol: RDEA3170 + Allopurinol | RDEA3170: RDEA3170 Alone | RDEA3170: RDEA3170 + Allopurinol
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12
hr | 1.06 [0.969 to 1.15] | 0.992 [0.890 to 1.10] | 43.2 [36.1 to 51.7] | 29.1 [23.9 to 35.4] | 11.5 [8.43 to 15.6] | 12.5 [8.99 to 17.4]

6. Primary Outcome: Amount Excreted in Urine as Unchanged Drug or Metabolite (Ae0-24)
Description: Ae0-24 of Allopurinol/Oxypurinol Alone and In Combination with RDEA3170
Time Frame: 22 days
Measure: Geometric Mean (95% Confidence Interval); unit: mg
Arm/Group | Allopurinol: Allopurinol Alone | Allopurinol: RDEA3170 + Allopurinol | Oxypurinol: Allopurinol Alone | Oxypurinol: RDEA3170 + Allopurinol
Number analyzed (Participants) | 12 | 12 | 12 | 12
mg | 25.4 [22.1 to 29.2] | 22.7 [19.2 to 26.9] | 231 [216 to 248] | 275 [262 to 290]
Statistical Analysis 1: Comparison: Allopurinol: Allopurinol Alone vs Allopurinol: RDEA3170 + Allopurinol; Test type: Non-Inferiority or Equivalence — Informal BE assessment using the conventional BE limits of 80% to 125%; Mixed Models Analysis; Fixed effect for treatment and random effects for subjects. GLMSRs are back-transformed to the original scale; Geometric Least Squares Mean Ratio (%) = 89.5, 90% CI 2-sided [81.8 to 98.0]
Statistical Analysis 2: Comparison: Oxypurinol: Allopurinol Alone vs Oxypurinol: RDEA3170 + Allopurinol; Test type: Non-Inferiority or Equivalence — Informal BE assessment using the conventional BE limits of 80% to 125%; Mixed Models Analysis; Fixed effect for treatment and random effects for subjects. GLMSRs are back-transformed to the original scale; Geometric Least Squares Mean Ratio (%) = 119, 90% CI 2-sided [114 to 125]

7. Primary Outcome: Renal Clearance of the Drug From Time Zero up to 24 Hours Postdose (CRL0-24)
Description: CLR0-24 of Allopurinol/Oxypurinol and RDEA3170 Alone and In Combination
Time Frame: 22 days
Measure: Geometric Mean (95% Confidence Interval); unit: mL/min
Arm/Group | Allopurinol: Allopurinol Alone | Allopurinol: RDEA3170 + Allopurinol | Oxypurinol: Allopurinol Alone | Oxypurinol: RDEA3170 + Allopurinol | RDEA3170: RDEA3170 Alone | RDEA3170: RDEA3170 + Allopurinol
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12
mL/min | 120 [106 to 135] | 103 [87.1 to 122] | 15.1 [13.0 to 17.6] | 29.2 [25.1 to 33.9] | 9.28 [7.43 to 11.6] | 9.75 [7.73 to 12.3]
Statistical Analysis 1: Comparison: Allopurinol: Allopurinol Alone vs Allopurinol: RDEA3170 + Allopurinol; Test type: Non-Inferiority or Equivalence — Informal BE assessment using the conventional BE limits of 80% to 125%; Mixed Models Analysis; Fixed effect for treatment and random effects for subjects. GLMSRs are back-transformed to the original scale; Geometric Least Squares Mean Ratio (%) = 87.5, 90% CI 2-sided [79.3 to 96.6]
Statistical Analysis 2: Comparison: Oxypurinol: Allopurinol Alone vs Oxypurinol: RDEA3170 + Allopurinol; Test type: Non-Inferiority or Equivalence — Informal BE assessment using the conventional BE limits of 80% to 125%; Mixed Models Analysis; Fixed effect for treatment and random effects for subjects. GLMSRs are back-transformed to the original scale; Geometric Least Squares Mean Ratio (%) = 193, 90% CI 2-sided [177 to 210]
Statistical Analysis 3: Comparison: RDEA3170: RDEA3170 Alone vs RDEA3170: RDEA3170 + Allopurinol; Test type: Non-Inferiority or Equivalence — Informal BE assessment using the conventional BE limits of 80% to 125%; Mixed Models Analysis; Fixed effect for treatment and random effects for subjects. GLMSRs are back-transformed to the original scale; Geometric Least Squares Mean Ratio (%) = 105, 90% CI 2-sided [94.4 to 117]

8. Primary Outcome: Pharmacodynamics (PD) Profile of Uric Acid From Serum and Urine
Time Frame: 22 days
Measure: Mean (Standard Error); unit: Percentage (%)
Arm/Group | RDEA3170: RDEA3170 Alone | Oxypurinol: RDEA3170 + Allopurinol | Allopurinol: Allopurinol Alone
Number analyzed (Participants) | 12 | 12 | 12
Percentage (%)
  Serum Urate Maximum % Change | -50.5 (2.43) [13.0 to 17.6] | -65.2 (1.57) [25.1 to 33.9] | -43.0 (1.57) [7.43 to 11.6]
  Urine Uric Acid % Change (0-24h) | 9.88 (7.61) | -21.6 (5.58) | -47.4 (2.67)
  Renal Clearance of Uric Acid % Change (0-24h) | 122 (46.8) | 125 (42.2) | -8.50 (6.04)
  Fract. Excretion of Uric Acid % Change (0-24h) | 77.4 (18.0) | 78.4 (21.9) | -12.0 (5.46)

9. Secondary Outcome: Incidence of Treatment-Emergent Adverse Events
Time Frame: 22 days
Measure: Number; unit: Number of participants
Arm/Group | RDEA3170: RDEA3170 Alone | Oxypurinol: RDEA3170 + Allopurinol | Allopurinol: Allopurinol Alone
Number analyzed (Participants) | 12 | 12 | 12
Number of participants | 2 (2.43) [13.0 to 17.6] | 1 (1.57) [25.1 to 33.9] | 3 (1.57) [7.43 to 11.6]

10. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: Cmax of RDEA3170 Alone and In Combination with Allopurinol
Time Frame: 22 days
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | RDEA3170: RDEA3170 Alone | RDEA3170: RDEA3170 + Allopurinol
Number analyzed (Participants) | 12 | 12
ng/mL | 14.6 [12.2 to 17.5] | 14.5 [11.7 to 17.9]
Statistical Analysis 1: Comparison: RDEA3170: RDEA3170 Alone vs RDEA3170: RDEA3170 + Allopurinol; Test type: Non-Inferiority or Equivalence — Informal BE assessment using the conventional BE limits of 80% to 125%; Mixed Models Analysis; Fixed effect for treatment and random effects for subjects. GLMSRs are back-transformed to the original scale; Geometric Least Squares Mean Ratio (%) = 98.7, 95% CI 2-sided [87.7 to 111]

11. Primary Outcome: Area Under the Concentration-time Curve From Time Zero up to 24 Hours Postdose (AUC 0-24)
Description: AUC 0-24 of RDEA3170 Alone and In Combination with Allopurinol
Time Frame: 22 days
Measure: Geometric Mean (95% Confidence Interval); unit: μg*hr/mL
Arm/Group | RDEA3170: RDEA3170 Alone | RDEA3170: RDEA3170 + Allopurinol
Number analyzed (Participants) | 12 | 12
μg*hr/mL | 120 [98.1 to 147] | 115 [96.5 to 137]
Statistical Analysis 1: Comparison: RDEA3170: RDEA3170 + Allopurinol; Test type: Non-Inferiority or Equivalence — Informal BE assessment using the conventional BE limits of 80% to 125%; Mixed Models Analysis; Fixed effect for treatment and random effects for subjects. GLMSRs are back-transformed to the original scale; Geometric Least Squares Mean Ratio (%) = 95.9, 95% CI 2-sided [88.4 to 104]

12. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to the Last Quantifiable Sampling Timepoint (AUC Last)
Description: AUC last of RDEA3170 Alone and In Combination with Allopurinol
Time Frame: 22 days
Measure: Geometric Mean (95% Confidence Interval); unit: ng·hr/mL
Arm/Group | RDEA3170: RDEA3170 Alone | RDEA3170: RDEA3170 + Allopurinol
Number analyzed (Participants) | 12 | 12
ng·hr/mL | 120 [98.1 to 147] | 115 [96.5 to 137]
Statistical Analysis 1: Comparison: RDEA3170: RDEA3170 Alone vs RDEA3170: RDEA3170 + Allopurinol; Test type: Non-Inferiority or Equivalence — Informal BE assessment using the conventional BE limits of 80% to 125%; Mixed Models Analysis; Fixed effect for treatment and random effects for subjects. GLMSRs are back-transformed to the original scale; Geometric Least Squares Mean Ratio (%) = 95.9, 95% CI 2-sided [88.4 to 104]

13. Primary Outcome: Amount Excreted in Urine as Unchanged Drug or Metabolite (Ae0-24)
Description: Ae0-24 of RDEA3170 Alone and In Combination with Allopurinol
Time Frame: 22 days
Measure: Geometric Mean (95% Confidence Interval); unit: ug
Arm/Group | RDEA3170: RDEA3170 Alone | RDEA3170: RDEA3170 + Allopurinol
Number analyzed (Participants) | 12 | 12
ug | 66.8 [51.8 to 86.1] | 67.2 [51.7 to 87.4]
Statistical Analysis 1: Comparison: RDEA3170: RDEA3170 Alone vs RDEA3170: RDEA3170 + Allopurinol; Test type: Non-Inferiority or Equivalence — Informal BE assessment using the conventional BE limits of 80% to 125%; Mixed Models Analysis; Fixed effect for treatment and random effects for subjects. GLMSRs are back-transformed to the original scale; Geometric Least Squares Mean Ratio (%) = 101, 95% CI 2-sided [86.7 to 117]

ADVERSE EVENTS:
Time Frame: 22 days
Description: Overall number of baseline participants used to determine number of participants at risk.
Groups:
- RDEA3170 10 mg qd: RDEA3170 10 mg qd
- RDEA3170 10 mg qd + Allopurinol 300 mg qd: RDEA3170 10 mg qd + Allopurinol 300 mg qd
- Allopurinol 300 mg qd: Allopurinol 300 mg qd
Arm/Group | RDEA3170 10 mg qd | RDEA3170 10 mg qd + Allopurinol 300 mg qd | Allopurinol 300 mg qd
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 2/12 | 1/12 | 3/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RDEA3170 10 mg qd (N=12) | RDEA3170 10 mg qd + Allopurinol 300 mg qd (N=12) | Allopurinol 300 mg qd (N=12)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall submit a copy of the Publication to Sponsor for review at least 45 days prior to its proposed submission. Sponsor reserves the right to delay any such publication for an additional period of 60 days. Upon Sponsor's request, PI agrees to delete from the proposed publication any Confidential Information. PI agrees not to release any publication without the prior written permission of Sponsor.